CLINICAL TRIAL: NCT01117506
Title: A Blood-based Gene Expression Test (Corus CAD or ASGES) for Obstructive Coronary Artery Disease Tested in Symptomatic Nondiabetic Patients Referred for Myocardial Perfusion Imaging.
Brief Title: Coronary Obstruction Detection by Molecular Personalized Gene Expression (Corus CAD or ASGES)
Acronym: COMPASS
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Collaborators: Cardiovascular Research Foundation, New York (Other); Piedmont Heart Institute, Inc., Atlanta, GA (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000007; COMPASS (Other: CardioDx)
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Chest Pain; Cardiovascular Diseases; Coronary Heart Disease; Angina Pectoris; CAD; CVD; CHD
Keywords: Angina Pectoris; Myocardial Ischemia; Molecular Genetics; Atherosclerosis; Corus CAD; ASGES; Age/Sex/Gene Expression Score; Gene Expression; GES; CAD; CVD; CHD; Precision Medicine; Clinical Validity; Myocardial Perfusion Imaging; Coronary Artery Disease; Chest Pain; Cardiovascular Disease; Coronary Heart Disease; MPI; COMPASS
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain; Cardiovascular Diseases; Coronary Disease; Angina Pectoris; Myocardial Ischemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA PAXgene
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Corus CAD (ASGES) — Age/Sex/Gene Expression Score - ASGES

SUMMARY:
To validate the use of Corus CAD (Age/Sex/Gene Expression score - ASGES) blood assay in subjects who are referred for the work-up of coronary artery disease. The study will evaluate the clinical utility of a gene expression test Corus CAD (Age, Sex, Gene Expression Score - ASGES) in subjects referred for myocardial perfusion imaging (MPI) work-up for suspected obstructive atherosclerotic coronary artery disease (CAD). The Corus CAD (ASGES) is a gene expression test that quantify the expression of multiple genes from circulating peripheral blood cells to detect the presence of clinically significant obstructive CAD in patients with chest pain.

DETAILED DESCRIPTION:
This prospective, multicenter study obtained peripheral blood samples for gene expression score (GES) before MPI in 537 consecutive patients Patients with abnormal MPI usually underwent invasive coronary angiography; all others had research coronary computed tomographic angiography, with core laboratories defining coronary anatomy A total of 431 patients completed GES, coronary imaging (invasive coronary angiography or computed tomographic angiography), and MPI Mean age was 56±10 years (48% women) The prespecified primary end point was GES receiver-operating characteristics analysis to discriminate ≥50% stenosis (15% prevalence by core laboratory analysis) Area under the receiver-operating characteristics curve for GES was 0 79 (95% confidence interval, 0 73-0 84; P<0 001), with sensitivity, specificity, and negative predictive value of 89%, 52%, and 96%, respectively, at a prespecified threshold of ≤15 with 46% of patients below this score The GES outperformed clinical factors by receiver-operating characteristics and reclassification analysis and showed significant correlation with maximum percent stenosis. Six-month follow-up on 97% of patients showed that 27 of 28 patients with adverse cardiovascular events or revascularization had GES >15 Site and core-laboratory MPI had areas under the curve of 0 59 and 0 63, respectively, significantly less than GES.

ELIGIBILITY:
Inclusion Criteria:

* Ages 45-90 for women; 35-90 for men.
* Stable chest pain syndrome (typical or atypical) or anginal equivalent in the judgment of the investigator (e.g., pain in the neck, jaw, arm or shoulder or dyspnea possibly due to cardiac ischemia).
* Referred for a stress test using MPI.
* The patient has signed the appropriate Institutional Review Board approved Informed Consent Form.

Exclusion Criteria:

* History of known MI or significant CAD.
* Current MI or acute coronary syndrome.
* Current New York Heart Association (NYHA) class III or IV congestive heart failure symptoms.
* Severe regurgitant or stenotic cardiac valvular lesion.
* Severe left ventricular systolic dysfunction (LVEF ≤ 35 % documented in the last year); if no assessment was performed or documented in the year preceding enrollment, presume normal LVEF.
* Active systemic infection (diagnosed by a combination of clinical symptoms and laboratory testing, including but not limited to fever, leukocytosis, positive blood cultures, pneumonia, urinary tract infection, or abscess in the preceding 2 months) or chronic infection (e.g., HIV, Hepatitis B or C, Tuberculosis).
* Protocol-specified rheumatologic, autoimmune or hematologic conditions (e.g., rheumatoid arthritis, systemic lupus erythematosis, polymyalgia rheumatica, or systemic sarcoidosis).
* Known or suspected diabetes mellitus or documented Hemoglobin A1c (HbA1c) ≥ 6.5; presume normal HbA1c if none documented.
* Total WBC ≥ 11,000 cells/ul and platelet count ≤ 75,000 cells/ul from a CBC with differential drawn within 7 days prior to enrollment [WBC ≥ 11,000 cells/ul and platelet count ≤ 75,000 cells/ul from a CBC drawn > 7 days prior need to be re-drawn at enrollment].
* Recipient of any organ transplant.
* Immunosuppressive or immunomodulatory therapy including any dose of systemic corticosteroids in the preceding 2 months.
* Chemotherapy in the preceding year.
* Major surgery in the preceding 2 months.
* Blood or blood product transfusion in the preceding 2 months.
* Subjects for whom all forms (stress or pharmacologic) of MPI are contraindicated.
* Subjects for whom invasive coronary angiography or coronary CT angiography is contraindicated, including IV beta-blocker.
* Subjects who planned to decline research CCTA or invasive coronary angiography, regardless of MPI result.
* Subjects with history of atrial fibrillation/flutter or frequent irregular or rapid heart rhythms.
* Known history of renal insufficiency (serum creatinine ≥ 2.0 mg/dL), or severe allergy to iodinated contrast.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll a patient population that presents with stable chest pain syndrome or anginal equivalent and referred for stress myocardial profusion imaging.
Sampling Method: Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy of Corus CAD (ASGES) in identifying the likelihood of obstructive CAD in a patient population with chest pain who are referred to a clinically-indicated myocardial profusion stress test. | Up to 45 days
  The primary endpoint for the COMPASS study is to assess whether the Corus CAD (ASGES) gene expression test performance is superior to an AUC of 0.5. The endpoint will be evaluated based on the current gold standard test for CAD, invasive coronary angiography, or a research CCTA after the subjects have undergone both the Corus CAD (ASGES) and MPI tests. Superiority will be assessed based upon demonstration of p<0.05 testing of the Corus CAD (ASGES) AUC versus an AUC of 0.50.

CONTACTS AND LOCATIONS:
Overall Officials: May Yau, MS, Study Director — CardioDx
Locations (7):
- United States (7):
  - Long Beach Memorial Hospital, Long Beach, California
  - Sutter Roseville Medical Center, Roseville, California
  - Pikes Peak Cardiology, Boulder, Colorado
  - Midwest Cardiology Associates, Overland Park, Kansas
  - St. Luke's Hospital, Kansas City, Missouri
  - Berks Cardiologists, Ltd, Wyomissing, Pennsylvania
  - Cardiovascular Associates of Virginia, Midlothian, Virginia

REFERENCES:
- [Result] Thomas GS, Voros S, McPherson JA, Lansky AJ, Winn ME, Bateman TM, Elashoff MR, Lieu HD, Johnson AM, Daniels SE, Ladapo JA, Phelps CE, Douglas PS, Rosenberg S. A blood-based gene expression test for obstructive coronary artery disease tested in symptomatic nondiabetic patients referred for myocardial perfusion imaging the COMPASS study. Circ Cardiovasc Genet. 2013 Apr;6(2):154-62. doi: 10.1161/CIRCGENETICS.112.964015. Epub 2013 Feb 15. PMID 23418288
- [Result] Voros S, Elashoff MR, Wingrove JA, Budoff MJ, Thomas GS, Rosenberg S. A peripheral blood gene expression score is associated with atherosclerotic Plaque Burden and Stenosis by cardiovascular CT-angiography: results from the PREDICT and COMPASS studies. Atherosclerosis. 2014 Mar;233(1):284-90. doi: 10.1016/j.atherosclerosis.2013.12.045. Epub 2014 Jan 20. PMID 24529158
- [Derived] Daniels SE, Beineke P, Rhees B, McPherson JA, Kraus WE, Thomas GS, Rosenberg S. Biological and analytical stability of a peripheral blood gene expression score for obstructive coronary artery disease in the PREDICT and COMPASS studies. J Cardiovasc Transl Res. 2014 Oct;7(7):615-22. doi: 10.1007/s12265-014-9583-3. Epub 2014 Aug 14. PMID 25119856